CLINICAL TRIAL: NCT02947919
Title: Impacto de la música en el estrés Preoperatorio en niños Sometidos a cirugía General
Brief Title: Impact of Music in the Preoperative Stress of Children Undergoing General Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with samples handling
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-242
Record Dates: First submitted 2016-10-13; First posted 2016-10-28 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Stress, Physiological; Stress, Psychological
Keywords: Perioperative Period; Music
MeSH Terms: conditions — Stress, Psychological | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Music in the perioperative period
  Interventions: Behavioral: Music
- Control (No Intervention): Usual treatment

INTERVENTIONS:
Behavioral: Music — A previously defined list of songs will be administered by headphones to these patients with an MP3 device with headphones.
  Arms: Intervention

SUMMARY:
Preoperative anxiety and stress are present in up to 60% of pediatric patients undergoing surgery, having a great physiological and emotional impact on children in both the short and long term. There are many reports on the use of music therapy in the perioperative period as a complementary technique in the preoperative stress and anxiety management. However, there are no assessments of the effect of this intervention on the physiological variables, such as salivary cortisol.

DETAILED DESCRIPTION:
60 patients aged 5-7 years, ASA (American Society of Anesthesiologists) status I-II, scheduled for general surgery at the Hospital of the Catholic University and associate institutions, will be considered for inclusion. 30 will receive music as intervention and 30 will received usual treatment. Salivary cortisol samples will be obtained preoperatively, in the surgical ward (OR), and in the post-anesthesia care unit (PACU). Secondary outcomes will be M-YPAS (Yale Preoperative Anxiety Scale) for children, and STAI (State-Trait Anxiety Inventory) for parents scales.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* ASA I-II
* Parents' consent

Exclusion Criteria:

* History of endocrine diseases (hypothyroidism, treatment with growth hormone, severely obese)
* Taking glucocorticoid inhalers or oral corticosteroids
* Children with severe hearing problems
* Patients requiring emergency surgery
* Refusal to participate in the study

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in salivary cortisol concentration | Before intervention (preoperative unit) and at an average of 30 minutes after surgery (at the post-anesthesia care unit)

SECONDARY OUTCOMES:
M-YPAS | Before intervention (preoperative unit) and at an average of 30 minutes after surgery (at the post-anesthesia care unit)
  M-YPAS (Yale Preoperative Anxiety Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo López, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Clinical Hospital - Pontificia Universidad Católica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCann ME, Kain ZN. The management of preoperative anxiety in children: an update. Anesth Analg. 2001 Jul;93(1):98-105. doi: 10.1097/00000539-200107000-00022. No abstract available. PMID 11429348
- [Background] Wennstrom B, Tornhage CJ, Nasic S, Hedelin H, Bergh I. The perioperative dialogue reduces postoperative stress in children undergoing day surgery as confirmed by salivary cortisol. Paediatr Anaesth. 2011 Oct;21(10):1058-65. doi: 10.1111/j.1460-9592.2011.03656.x. Epub 2011 Jul 20. PMID 21771174